CLINICAL TRIAL: NCT03160924
Title: The Impact of Enhanced Recovery After Surgery (ERAS) Program on Clinical and Immunological Outcomes for Minimally-invasive Gastrectomy: A Randomized Controlled Trial
Brief Title: The Impact of Enhanced Recovery After Surgery (ERAS) Program on Clinical and Immunological Outcomes for Minimally-invasive Gastrectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHAN SHANNON MELISSA, Resident Specialist, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CRE2015.530
Record Dates: First submitted 2017-05-15; First posted 2017-05-19 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Enhanced Recovery After Surgery for Laparoscopic Gastrectomy for Patients With Gastric Cancer
Keywords: Enhanced recovery after surgery; ERAS; Fast track recovery; Laparoscopic gastrectomy; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Intervention Model Description: This is a randomised controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Recovery After Surgery (ERAS) (Active Comparator): In this arm, the ERAS perioperative care program will be applied.
  1. Preoperative counselling by surgeon, dietician and physiotherapist
  2. Preoperative carbohydrate-loaded drink 800ml 12.5% Carbohydrate drink 8h before surgery 400ml 12.5% Carbohydrate drink 4h before surgery (Omit 4h drink if patient has DM)
  3. Fluid restriction, avoid opioids, use of Cox-II inhibitors as analgesics
  4. Avoid use of drains
  5. Early resumption of diet
  6. Early mobilisation with physiotherapist
  7. Dietary counselling by dietician
  8. Early discharge if fulfil discharge criteria.
  Discharge criteria:
  Adequate pain control with oral analgesics Ability to tolerate soft diet Passage of flatus Mobilization
  Patients will be called by doctors every day after discharge to monitor their clinical status. There will be a low threshold for readmitting patients. Patients will also be given a hotline to call if they feel unwell. They will be seen in clinic on post-operative D7 and D14.
  Interventions: Other: Enhanced Recovery After Surgery (ERAS)
- Conventional perioperative program (No Intervention): In this arm, the conventional preoperative program will be applied.
  1. No preoperative counselling
  2. No Preoperative carbohydrate-loaded drink
  3. Routine anaesthesia, no specific protocol on fluid restriction, opioids will be used as usual. Tramadol would be used as postoperative pain control.
  4. Routine use of drains
  5. Diet will be resumed when there is flatus clinically
  6. Mobilisation as per patient's wish
  7. Dietary counselling by dietician
  8. Discharge if fulfil discharge criteria.
  Discharge criteria:
  Adequate pain control with oral analgesics Ability to tolerate soft diet Passage of flatus Mobilization
  Patients will be seen in clinic on post-operative D14.

INTERVENTIONS:
Other: Enhanced Recovery After Surgery (ERAS) — same as above as described in the "arms".
  Arms: Enhanced Recovery After Surgery (ERAS)

SUMMARY:
Over the past two decades, fast track surgery, also known as "enhanced recovery after surgery (ERAS)" has been initiated and developed in colorectal surgery by Kehlet. The program is rapidly gaining popularity due to the significant benefits demonstrated in lowering complication rates and reducing hospital stay and costs. The benefits demonstrated in colorectal surgery by randomized trials and meta-analyses reduced pain, morbidity and hospital stay. Data in gastrectomy however, is scarce. Therefore the aim of this study is to compare the outcomes of laparoscopic gastrectomies with two different perioperative approaches, the traditional and the ERAS approach in a setting of a randomised controlled trial.

DETAILED DESCRIPTION:
Over the past two decades, fast track surgery, also known as "enhanced recovery after surgery (ERAS)" has been initiated and developed in colorectal surgery by Kehlet. The program is rapidly gaining popularity due to the significant benefits demonstrated in lowering complication rates and reducing hospital stay and costs. The benefits demonstrated in colorectal surgery by randomized trials and meta-analyses reduced pain, morbidity and hospital stay. Data in gastrectomy however, is scarce. Therefore the aim of this study is to compare the outcomes of laparoscopic gastrectomies with two different perioperative approaches, the traditional and the ERAS approach in a setting of a randomised controlled trial.

ERAS involves an integrated multi-disciplinary program of various medical interventions involving surgeons, anaesthetists, physiotherapists, dieticians and nurses, aiming at enhancing postoperative recovery by reducing surgical stress response resulting in earlier discharge and potentially reduced morbidities. The program focuses on minimising the impact of surgery on patients' homeostasis. The reduction of postoperative physiological stress by the attenuation of the neurohormonal response to the surgical intervention not only provides the basis for a faster recovery, but also diminishes the risk of organ dysfunction and complications. The ERAS program consists of well-organised pathways of clinical interventions that begin from out-patient preoperative information, counselling and physical optimization, proceeding to pre-, intra- and postoperative protocol-driven actions and end with patient discharge following pre-established criteria. The main pillars of ERAS program consist of extensive preoperative counselling, non sedative premedication, no preoperative fasting but with pre-operative carbohydrate loading, tailored anaesthesiology, peri-operative intravenous fluid restriction, non-opioid pain management, non routine use of nasogastric tubes, early removal of urinary catheter, and early postoperative feeding and mobilization.

ERAS program will be implemented in one arm and the other arm would be conventional peri-operative care. This is a randomised controlled study. Apart from clinical outcomes, the immunological outcomes will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive patients undergoing elective gastrectomy with the minimally-invasive approach
2. Aged between 18 and 75 years
3. American Society of Anesthesiologists (ASA) grading I-II
4. No severe physical disability
5. Patients who require no assistance with the activities of daily living
6. Informed consent available.

Exclusion Criteria:

1. Preoperative chemotherapy or radiotherapy
2. Known metastatic disease
3. Previous history of midline laparotomy
4. Gastric outlet obstruction
5. Known immunological dysfunction (e.g. HIV infection)
6. Patients on steroids or immunosuppressive agents, patients with chronic pain syndrome and patients with chronic renal or liver disease
7. Patients who are pregnant and mentally incapable of consent

Post-randomization exclusion criteria:

Since the operation itself is a determinant to postoperative course and management, the withdrawal criteria were established as follows:

1. Intraoperative blood loss >= 500ml
2. Prolonged operation >6hrs
3. Gastrectomy not proceeded due to presence of peritoneal metastasis Concomitant resection of organs other than the gallbladder, eg. spleen, bowel

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Post-operative hospital stay | Within 30 days
  The number of days patient stays in hospital after the surgery

SECONDARY OUTCOMES:
Serum lymphocyte counts | Within 5 days of the surgery
  This is used to assess the patient's immunological status after the surgery.
Post-operative pain scores | Within 2 weeks
  Pain scores on visual analogue scale (from 0 that implies no pain at all, to 100 which implies the worst pain imaginable) assessed daily from day 0 onwards till discharge. Pain assessments will be conducted after patients have been in a resting supine position for 5 minutes and then repeated after coughing for ten times.
Forced vital capacity | Within 2 weeks
  This will be done in terms of peak flow rate at bedside.
Mortality and morbidity | Within 30 days
  The morbidities would be recorded according to predefined criterion. Mortalities within 30 days would be included.
Readmission rate | Within 30 days
  Readmission of more than 24 hours would be counted as readmission
Quality of life assessments | within 4 weeks
  This will be measured by European organisation for Research and Treatment of Cancer (EORTC)-stomach questionnaires
Direct hospital costs | within 30days
  All costs involving the admission and readmissions

CONTACTS AND LOCATIONS:
Overall Officials: Shannon M Chan, MBCHB, FRCS, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese Universtiy of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The data of the patients will only be available to researches participating in this study.